CLINICAL TRIAL: NCT01873326
Title: Randomized Phase II Trial of Paclitaxel, Ifosfamide and Cisplatin (TIP) Versus Bleomycin, Etoposide and Cisplatin (BEP) for Patients With Previously Untreated Intermediate- and Poor-Risk Germ Cell Tumors
Brief Title: Paclitaxel, Ifosfamide and Cisplatin (TIP) Versus Bleomycin, Etoposide and Cisplatin (BEP) for Patients With Previously Untreated Intermediate- and Poor-risk Germ Cell Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Southern California (Other); Mayo Clinic (Other); University of Pittsburgh (Other); University of North Carolina (Other); University of Chicago (Other); Stanford University (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-074
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Germ Cell Tumors
Keywords: newly diagnosed GCT; Intermediate; Poor-Risk; BLEOMYCIN; CISPLATIN; ETOPOSIDE (VP-16); IFOSFAMIDE; TAXOL (PACLITAXEL); 13-074
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Paclitaxel; Ifosfamide; Cisplatin; Mesna; Bleomycin; Etoposide

ARMS (2):
- Paclitaxel, Ifosfamide and Cisplatin (TIP) (Experimental): Paclitaxel 120 mg/m2 IV over 120-180 min Days 1 and 2 (+/- 4 days)* Mesna 120 mg/m2 IV (duration of infusion per institutional guidelines) approximately 30 minutes prior to initiation of ifosfamide Days 1-5 (+/- 4 days)* Ifosfamide 1200 mg/m2 IV over approximately 60 to 120 min Days 1-5 or per institutional guidelines (mixed 1:1 with mesna) (+/- 4 days)* Mesna** 1200 mg/m2 IV over approximately 60-120 min or per institutional guidelines (mixed 1:1 with ifosfamide)(+/- 4 days)* Cisplatin 20 mg/m2 IV over approximately 30 min Days 1-5 (+/- 4 days)*
  **Additional mesna may be given at the discretion of the investigator
  *Paclitaxel or Ifosfamide or Mesna or Cisplatin or any combination of these agents can be held as needed for patient safety on a given day between days 1-5 but must be made up within 4 days to avoid a protocol violation.
  Interventions: Drug: Paclitaxel; Drug: Ifosfamide; Drug: Cisplatin; Drug: Mesna
- Bleomycin, Etoposide and Cisplatin (BEP) (Active Comparator): Cisplatin 20 mg/m2 IV over approximately 30 min Days 1-5 (+/- 4 days)* Etoposide 100 mg/m2 IV over approximately 1 hour Days 1-5 (+/- 4 days)* Bleomycin 30 U flat dose IV push Days 2, 8 and 15 (all +/- 4 days)
  *Etoposide or Cisplatin or both can be held as needed for patient safety on a given day between days 1-5 but must be made up within 4 days to avoid a protocol violation.
  Interventions: Drug: Cisplatin; Drug: Bleomycin; Drug: Etoposide

INTERVENTIONS:
Drug: Paclitaxel
  Arms: Paclitaxel, Ifosfamide and Cisplatin (TIP)
Drug: Ifosfamide
  Arms: Paclitaxel, Ifosfamide and Cisplatin (TIP)
Drug: Cisplatin
Drug: Mesna
  Arms: Paclitaxel, Ifosfamide and Cisplatin (TIP)
Drug: Bleomycin
  Arms: Bleomycin, Etoposide and Cisplatin (BEP)
Drug: Etoposide
  Arms: Bleomycin, Etoposide and Cisplatin (BEP)

SUMMARY:
The purpose of this study is to learn about the safety and effectiveness of two different drug combinations in patients who have intermediate- and poor-risk germ cell tumors (GCT). One combination of drugs, paclitaxel, ifosfamide and cisplatin (TIP), is experimental. The other combination of drugs, bleomycin, etoposide and cisplatin (BEP), is the standard of care treatment for intermediate- and poor-risk germ cell tumors. However, BEP does not cure every patient and therefore newer treatments are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Patients with newly diagnosed GCT
* Pathology confirmation of GCT histology at MSKCC or a collaborating treating institution. In exceptional circumstances, patients without pathological diagnosis may be included in the study following discussion with the national principal investigator, Dr. Feldman,(or national Co-PI or MSKCC Co-PI if the national PI is unavailable) if they meet the one of the following criteria:
* Patients with a testicular mass (detected clinically and/or by ultrasound), and/or mediastinal or retroperitoneal lymphadenopathy or pineal tumor AND elevated serum tumor markers (HCG and/or AFP). Patients with elevated LDH only will not be included without pathological confirmation of GCT since LDH is a nonspecific marker for GCT and could potentially be elevated in other malignancies such as lymphomas.

This is because patients may present with a clinical scenario consistent with GCT (elevated serum tumor markers, testicular mass and retroperitoneal lymphadenopathy) with a concurrent life-threatening oncologic emergency that require immediate treatment. In this case, initial treatment without biopsy confirmation is usually recommended and tissue confirmation may be obtained after initiating therapy.

* Patients must have measurable or evaluable disease.
* Patients must be classified as having intermediate or poor-risk germ cell tumor, as follows:

  * Intermediate-risk (Modified*) a) Testis or retroperitoneal primary NSGCT with lymph node and/or lung metastasis but without non-pulmonary visceral metastasis AND any of the following pretreatment serum tumor marker (STM) values: i. Lactate dehydrogenase (LDH) from 3 to <10 x ULN (*This differs from the original IGCCCG criteria which includes patients with LDH from 1.5 to 10 x ULN).

ii. Serum human chorionic gonadotrophin (HCG) from 5,000 to < 50,000 MIU/mL iii. Serum alpha-fetoprotein (AFP) from 1,000 to <10,000 ng/mL b) Seminoma histology regardless the primary site or serum tumor markers with any non-pulmonary visceral metastasis (liver, bone, brain, etc).

* Poor-risk (any of the following):

  1. Testis or retroperitoneal NSGCT primary with non-pulmonary visceral metastasis (liver, bone, brain, etc) regardless the STM values.
  2. Mediastinal NSGCT primary site of disease regardless the presence/absence of visceral metastasis or STM values.
  3. Testis or retroperitoneal NSGCT primary without non-pulmonary visceral metastasis but with poor-risk STM values:
* i. LDH ≥ 10 x ULN
* ii. HCG ≥ 50,000 MIU/mL
* iii. AFP ≥ 10,000 ng/mL

  * Patients who received prior radiation therapy (RT) for treatment of germ cell tumor are eligible for this study as long as there is evidence of progressive disease determined by tumor markers or other sites of metastases outside of the radiated site. Radiation must be completed prior to starting chemotherapy with the exception of brain metastases where chemotherapy and radiation can be given concurrently. Toxicity from radiation must have recovered to grade 1 or less prior to initiating chemotherapy.
  * Patients must have recovered from prior surgery based on treating physician's discretion.
  * Patients of reproductive potential must agree to use effective contraception during the period of therapy
  * Signed informed consent.
  * Diffusion lung capacity for carbon monoxide (DLCO) adjusted for hemoglobin ≥60% predicted, except if related to high volume metastatic GCT to the lungs in which case there is no minimum DLCO requirement. In some cases, patients may not be able to undergo PFT testing due to the severity of their presentation. such as those with high volume lung metastases or tumor-related pain (from large mediastinal masses, pleural disease, etc.) limiting their ability to complete PFTs. Even when PFTs can be completed in these cases, patients will still be eligible if the low DLCO can be attributed directly to the patient's disease (e.g., large mediastinal mass) rather than intrinsic lung disease. Since there is no minimum DLCO for these patients, under these extraordinary circumstances, this will be allowed. Most patients in this situation will be expected to receive disease-stabilizing chemotherapy. An unadjusted DLCO may be used in place of the DLCO adjusted for hemoglobin in certain situations as per institutional policy. For example, MSKCC policy is to not adjust the DLCO for hemoglobin when the hemoglobin is ≥ 14.6 g/dL for males and ≥ 13.4 g/dL for females. In these cases, the unadjusted DLCO must be >60% predicted.
* Laboratory criteria for protocol entry (obtained ≤ 14 days before initiation of therapy):
* WBC ≥ 3000/UL and Platelet count ≥ 100,000/UL
* Serum creatinine ≤ 1.5 mg/dL or estimated GFR (by Cockcroft-Gault) ≥50mL/min or 12 or 24 hour urine creatinine clearance ≥ 50 mL/min, unless renal insufficiency is due to tumoral ureteral obstruction in which case eligibility will be determined by national the principal investigator (or national co-PI or MSKCC co-PI if the national PI is unavailable) with notification of the MSKCC IRB.
* AST/ALT ≤ 3 x ULN and total bilirubin ≤ 2.0 x ULN. In the setting of metastatic disease to the liver, AST/ALT may be ≤5x ULN and total bilirubin ≤2.5 x ULN. If a patient is known or suspected to have Gilbert's disease, total bilirubin up to ≤2.5 x ULN is allowed.

Exclusion Criteria:

* Any prior chemotherapy. The only exception will be patients with a history of stage I seminoma treated with adjuvant carboplatin for 1 or 2 cycles.
* Concurrent treatment with any cytotoxic therapy.
* Known concurrent malignancy (except for non-melanoma skin cancer).
* Patients known to be HIV positive and receiving HAART.
* Presence of an active infection. Patients with fever assessed to be "tumor fever" but without active evidence of infection (e.g. blood cultures are negative) are eligible. In addition, patients who have an infection but without evidence of fever for 48 hours on antibiotics will be eligible.
* Inability to comply with the treatment protocol or to undergo prespecified follow-up tests for safety or effectiveness.
* Pregnant patients are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
favorable best response rate | 6 months
  Favorable best response is defined as complete response or partial response with negative tumor markers. Patients will be considered evaluable for the primary endpoint of favorable response within the first 6 months if they complete at least 3 cycles of study treatment (without switch to an alternative chemotherapy regimen) and achieve a confirmed partial response with negative markers or confirmed complete response (considered as favorable responses). Patients will also be considered evaluable for the primary endpoint if they develop disease progression during the treatment portion of the study regardless of how many cycles of chemotherapy they received or if they achieve an incomplete response after completion of study treatment (considered as not having a favorable response)."

SECONDARY OUTCOMES:
overall best response | 3 years
  Overall best response refers to the best response achieved by a patient to either TIP or BEP over the course of the entire study.
progression-free survival (PFS) | 3 years
  Progression-free survival (PFS) will be calculated from the date of treatment start until disease progression, death, or last followup, whichever comes first. The following are included as PFS events: incomplete response (IR), relapse or disease progression, and death.
overall survival (OS) | 3 years
  Overall survival will be calculated from the date of treatment start until death, regardless of the cause.
toxicity | 30 days after completion of the last cycle of chemotherapy.
  Toxicity will be assessed based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade of each toxicity will be recorded for each patient over the course of treatment (all cycles). Special emphasis will be placed on comparisons of the frequency of Grade 3/4 toxicities between the TIP and BEP arms.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (13):
- United States (13):
  - University of Southern California, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Follow-up Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/